CLINICAL TRIAL: NCT04771754
Title: The Effect of Dolutegravir on Whole-body Insulin Sensitivity, Lipid and Endocrine Profile in Healthy Volunteers
Acronym: DTG Clamp
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CRF003
Record Dates: First submitted 2021-01-20; First posted 2021-02-25 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: HIV-1-infection on Healthy Volunteers
Keywords: HIV; Dolutegravir; Insulin
MeSH Terms: conditions — Insulin Resistance | interventions — dolutegravir

STUDY DESIGN:
Intervention Model Description: Subjects will be randomised to start on dolutegravir 50 mg once daily OR no treatment for the first 28 day dosing phase of the study then will cross over to the alternative for the second dosing phase, following a 2 week washout period (equivalent to 5+ dolutegravir elimination half-lives).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): * Dolutegravir - 50 mg once daily, orally administered for the first 28 days of the study.
  * No treatment for the last 44 days of the study.
  Interventions: Drug: Dolutegravir
- Arm 2 (Experimental): * No treatment for the first 28 days of the study.
  * Dolutegravir - 50 mg once daily, orally administered for the last 28 days of the study (day 44-72).
  Interventions: Drug: Dolutegravir

INTERVENTIONS:
Drug: Dolutegravir — 50 mg once daily orally
  Other Names: Tivicay

SUMMARY:
This study will investigate changes in insulin resistance, lipid metabolism and endocrine profile in HIV-negative subjects exposed to dolutegravir (an antiretroviral drug used in HIV treatment) in order to investigate the role all these different factors may potentially have in weight gain recently reported in clinical cohorts.

DETAILED DESCRIPTION:
A randomised, crossover study investigating the difference in changes in insulin sensitivity (determined by peripheral glucose uptake using a euglycaemic clamp) with the administration of dolutegravir (DTG) compared to no DTG for 28 days in HIV seronegative healthy volunteers.

Participants will be randomised 1:1 to one of two arms:

Group 1:

* Dolutegravir 50 mg once daily for the first 28 days of the study.
* No treatment for the last 44 days of the study.

Group 2:

* No treatment for the first 28 days of the study.
* Dolutegravir 50 mg once daily for the last 28 days of the study (day 44-72).

Research bloods, endocrine profiles, weight and urine samples will be collected at baseline, as well as day 28, 44, and 72 to enable comparative analyses.

Participants will be closely monitored whilst taking the study medications. Participants will exit the study 72 days post-randomisation, with a follow-up call 28 days after exiting.

ELIGIBILITY:
Inclusion Criteria

* Willing and able to provide informed consent
* Cis-Male and Cis-Female healthy subjects without underlying conditions
* Subjects must have documented negative HIV serology by ELISA and P24 antigen and not receiving anti-HIV pre-exposure prophylaxis (PreP)
* Subjects must be clinically well volunteers aged between 18 to 60 years with BMI <30 kg/m2 but >18 kg/m2
* Healthy, as determined by the investigator or medically qualified designee based on a medical evaluation, including medical history, physical examination, laboratory tests, and cardiac evaluation (including ECG)
* Non-fasting blood glucose, total cholesterol and triglycerides within normal limits
* Subjects should have complete blood count (FBC) with normal differential and platelet count (detail below of specified normal range, table 1)

Table 1 - Compete FBC with normal differential & platelets count ranges Test Male Normal Range Female Normal Range Haemoglobin (g/L) 130-168 114-150 White blood cell count (x109/L) 4.2-10.6 4.2-11.2 Neutrophil count (x109/L) 2.0 - 7.1 Lymphocyte count (x109/L) 1.1 - 3.6 Monocyte count (x109/L) 0.2 - 0.9 Eosinophil count (x109/L) 0.0 - 0.5 Basophil count (x109/L) 0.0 - 0.2

* A female, may be eligible to enter and participate in the study if she:

  * is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or,
  * is of child-bearing potential with a negative pregnancy test at both Screening and Day 1 and agrees to use one of the following methods of contraception to avoid pregnancy:
  * Complete abstinence from penile-vaginal intercourse. Abstinence is acceptable only as true abstinence when this is in line with the preferred and usual lifestyle of the participant;
  * Any intrauterine device with published data showing that the expected failure rate is <1% per year (not all intrauterine devices meet this criterion, see Appendix 6] for an example listing of approved intrauterine devices);
  * Male partner sterilization confirmed prior to the female subject's entry into the study, and this male is the sole partner for that subject;
  * Approved hormonal contraception (see Appendix 6] for a listing of examples of approved hormonal contraception)*;
  * Any other method with published data showing that the expected failure rate is <1% per year
* Men who have partners who are women of childbearing potential (WOCBP - definition in Appendix 6) must be using an adequate method of contraception to avoid pregnancy in their partner throughout the study and for a period of at least 4 weeks after the study;
* Complete abstinence from penile-vaginal intercourse. Abstinence is acceptable only as true abstinence when this is in line with the preferred and usual lifestyle of the patient;
* Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide);
* Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion, see Appendix 4 for an example listing of approved IUDs) plus male condom;
* Sterilisation confirmed prior to the subject's entry into the study
* Approved hormonal contraception used by female partner (see protocol appendix 4 for a listing of examples of approved hormonal contraception) plus male condom;
* Any other method with published data showing that the expected failure rate is <1% per year and not containing hormones plus male condom.
* Any contraception method must be used consistently, in accordance with the approved product label and for at least four weeks after discontinuation of IMP (Appendix 6).

Any contraception method must be used consistently, in accordance with the approved product label and for at least 28 days prior to the first dose of study medication and 4 weeks after discontinuing the study medication.

4.1.2 Exclusion Criteria

* Subjects with a waist hip ratio > 0.97 or BMI > 30kg/m2 and BMI <18 kg/m2 will be excluded
* Acute or chronic hepatitis B infection (determined by positive hepatitis B surface antigen result at the screening visit)
* Acute or chronic hepatitis C infection (determined by positive hepatitis C antibody result at the screening visit)
* Diabetes mellitus, other metabolic syndrome or disease process in the opinion of the investigator likely to cause marked disturbance in glucose and lipid homeostasis including hypertension. Subject with HbA1c >42 mmol/mol will be excluded.
* History or presence of allergy to the dolutegravir
* ALT or AST greater than or equal to 1.5 x Upper Limit of Normal (ULN) and total bilirubin greater than or equal to 1.5 x ULN excluded;
* Pregnancy and breastfeeding women
* Alcohol consumption >10 units/week
* Clinically relevant drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study.
* Unable to refrain from the use of prescription (e.g., dofetilide) or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives prior to the baseline visit and throughout the study until the follow-up period, unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise participant safety.
* This includes on-going therapy with any of the following

  * Metabolically active medications
  * Any lipid-lowering medication
  * Any testosterones treatments or supplements - Glucocorticoids including inhaled steroids except for 'as necessary' use
  * Beta-blockers
  * Thiazide diuretics and indapamide
  * Thyroid preparations
  * Psychotropic agents
  * Anabolic steroids
  * Megestrol acetate
  * Dofetilide (or pilsicainide)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Bryne, Principal Investigator — Chelsea and Westminster Hospital
Locations (1):
- Arnold Xhikola, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: * Dolutegravir - 50 mg once daily, orally administered for the first 28 days of the study.
  * No treatment for the last 44 days of the study.
  Dolutegravir: 50 mg once daily orally
- Arm 2: * No treatment for the first 28 days of the study.
  * Dolutegravir - 50 mg once daily, orally administered for the last 28 days of the study (day 44-72).
  Dolutegravir: 50 mg once daily orally
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 8 | 8
Completed | 7 | 8
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants] — Population: Participant lost to follow up/ dropout
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 7 | 8 | 15
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Sensitivity in Participants From Baseline to End of Study Between Two Crossover Groups.
Description: Change in insulin sensitivity will be determined by peripheral glucose uptake using a euglycaemic clamp.
Time Frame: Baseline, day 28 and 72 for both groups.
Population: Dolutegravir versus No Treatment Two sample Wilcoxon rank sum (Mann Whitney) test
Measure: Mean (Standard Deviation); unit: (mg/kg/min)
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 7 | 8
(mg/kg/min)
  Baseline | 7.749985 (3.520332) | 6.286017 (2.072026)
  Day 28 | 8.716221 (2.600469) | 6.815305 (2.404083)
  Day 72: number analyzed (Participants) | 6 | 8
  Day 72 | 10.62598 (5.250227) | 7.684051 (2.516086)

2. Secondary Outcome: Effect of Dolutegravir on Adipocytokines.
Description: Fasting adiponectin levels in blood.
Time Frame: Baseline, day 28 and 72 for both groups.
Population: Dolutegravir versus No Treatment Two sample Wilcoxon rank sum (Mann Whitney) test
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 7 | 8
ng/mL
  Adiponectin Baseline | 7066.733 (4002.151) | 7555.781 (4201.587)
  Adiponectin Day 28 | 7573.153 (4832.789) | 8294.638 (5464.168)
  Adiponectin Day 72 | 6531.739 (3687.814) | 9220.179 (5437.189)

3. Secondary Outcome: Effect of Dolutegravir on Pituitary Hormones
Description: Cortisol
Time Frame: Baseline, day 28 and 72 for both groups.
Measure: Mean (Standard Deviation); unit: nmol /L
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 7 | 8
nmol /L
  Baseline | 229.7143 (106.6173) | 307.25 (116.4643)
  Day 28 | 290.8571 (116.7325) | 304 (102.0868)
  Day 72 | 233.375 (102.841) | 272.8889 (116.7994)

4. Secondary Outcome: Effect of Dolutegravir on Changes in Indirect Calorimetry
Description: Indirect calorimetry by ventilated hood expires gas analysis will be used to determine energy expenditure during the course of the clamp procedures.
Time Frame: Baseline, day 28 and 72 for both groups.
Reporting Status: Not Posted

5. Secondary Outcome: Effect of Dolutegravir on Adipocytokines.
Description: Fasting Leptin levels in blood.
Time Frame: Baseline, day 28 & 72 for both groups.
Population: Dolutegravir versus No Treatment Two sample Wilcoxon rank sum (Mann Whitney) test
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 7 | 8
ug/L
  Leptin Baseline | 8.687143 (5.559331) | 12.58571 (11.13826)
  Leptin Day 28 | 12.16571 (10.39278) | 10.57286 (8.23104)
  Leptin Day 72 | 13.768 (8.141939) | 12.22 (9.240835)

6. Secondary Outcome: Effect of Dolutegravir on Adipocytokines.
Description: Fasting Ghrelin levels in blood.
Time Frame: Baseline, day 28 & 72 for both groups.
Population: Dolutegravir versus No Treatment Two sample Wilcoxon rank sum (Mann Whitney) test
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 7 | 8
ng/L
  Ghrelin Baseline | 3555.059 (2749.332) | 3873.6 (2962.185)
  Ghrelin Day 28 | 1873.901 (1817.324) | 4171.744 (1671.54)
  Ghrelin Day 72 | 4557.219 (4493.846) | 2826.041 (2823.855)

7. Secondary Outcome: Effect of Dolutegravir on Pituitary Hormones
Description: Prolactin
Time Frame: Baseline, day 28 and 72 for both groups.
Measure: Mean (Standard Deviation); unit: mIU /L
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 7 | 8
mIU /L
  Baseline | 261 (117.5131) | 196.625 (54.52113)
  Day 28 | 173.7143 (110.7019) | 231.5 (138.0497)
  Day 72 | 238.5 (112.5052) | 227.1111 (86.96327)

8. Secondary Outcome: Effect of Dolutegravir on Pituitary Hormones
Description: Luteinsing Hormone Level
Time Frame: Baseline, day 28 and 72 for both groups.
Measure: Mean (Standard Deviation); unit: mIU /L
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 7 | 8
mIU /L
  Baseline | 4.585714 (5.440107) | 2.1625 (0.8667468)
  Day 28 | 3.171429 (1.900626) | 2.825 (0.9852483)
  Day 72 | 2.4 (1.656157) | 2.355556 (1.35904)

9. Secondary Outcome: Effect of Dolutegravir on Pituitary Hormones
Description: Growth Hormone
Time Frame: Baseline, day 28 and 72 for both groups.
Measure: Mean (Standard Deviation); unit: μg /L
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 7 | 8
μg /L
  Baseline | 0.1642857 (0.1137039) | 0.15875 (0.1211183)
  Day 28 | 1.144286 (2.545361) | 0.85 (1.859416)
  Day 72 | 0.58375 (1.241818) | 0.3322222 (0.6257551)

10. Secondary Outcome: Effect of Dolutegravir on Lipid Profile Including Lipid Fractions
Description: Total Cholesterol
Time Frame: Baseline, day 28 and 72 for both groups.
Measure: Mean (Standard Deviation); unit: mmol /L
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 7 | 8
mmol /L
  Baseline | 4.071429 (0.3638419) | 4.25 (0.8244305)
  Day 28 | 3.681429 (1.076358) | 4.165 (0.5593619)
  Day 72 | 2.965 (1.397252) | 3.867778 (1.775414)

11. Secondary Outcome: Effect of Dolutegravir on Lipid Profile Including Lipid Fractions
Description: Triglycerides
Time Frame: Baseline, day 28 and 72 for both groups.
Measure: Mean (Standard Deviation); unit: mmol /L
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 7 | 8
mmol /L
  Baseline | 0.7214286 (0.310023) | 0.87 (2186974)
  Day 28 | 0.8342857 (0.3867754) | 0.76 (0.1962506)
  Day 72 | 0.62375 (0.4254388) | 0.6355556 (0.3005458)

12. Secondary Outcome: Changes in Food Intake by Food Preference Questionnaire
Description: Changes in food intake Food preference questionnaire for adolescents and adults (FPQ)
  1- Scoring of Individual Items
  Each food item is rated on a 5-point Likert scale:
  1. = Dislike a lot
  2. = Dislike a little
  3. = Neither like nor dislike
  4. = Like a little
  5. = Like a lot
  Responses marked as "Not applicable" are treated as missing and not included in scoring.
  Food Category Scores
  Items are grouped into six categories, each scored by averaging across the foods in that group:
  Vegetables (18 items)
  Fruits (7 items)
  Meat/Fish (12 items)
  Dairy (10 items)
  Snacks (9 items)
  Starches (6 items)
  The category score is the mean of item scores in that category (sum ÷ number of items).
  For both individual items and category scores:
  Minimum possible score = 1 ("Dislike a lot") Maximum possible score = 5 ("Like a lot")
  Direction of Scoring On the FPQ, higher scores reflect greater liking of the foods, Lower scores indicate less liking.
  'scores on a scale'
Time Frame: Baseline, day 28 and 72 for both groups.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 7 | 8
scores on a scale
  Baseline | 3.719047619 (0.464914105) | 4.0375 (0.458087055)
  Day 28 | 3.654285714 (0.434338447) | 4.066666667 (0.339461379)
  Day 72 | 3.726428571 (0.44250229) | 3.983958333 (0.561874305)

13. Secondary Outcome: Change in Sleep Parameters by Sleep Questionnaires
Description: changes in sleep parameters by Pittsbrough Sleep Quality Index (PSQI)
  1. Scoring Components
     The PSQI has 19 self-rated items, grouped into 7 component scores:
     Subjective sleep quality
     Sleep latency
     Sleep duration
     Habitual sleep efficiency
     Sleep disturbances
     Use of sleeping medication
     Daytime dysfunction
     Each component is scored from 0 to 3, where higher values indicate worse sleep in that domain.
  2. Global Score
  The 7 component scores are summed to yield a global PSQI score ranging from 0 to 21.
  0 = no difficulty / very good sleep quality
  21 = severe difficulties / very poor sleep quality
  3- Interpretation
  A global score > 5 is commonly used as a cut-off to distinguish between "good sleepers" (≤5) and "poor sleepers" (>5).
  4- Direction of Scoring
  On the PSQI, higher scores indicate worse outcomes (poorer sleep quality).
  Lower scores indicate better sleep quality.
  Unit of Measue = Score on a scale
Time Frame: Baseline, day 28 and 72 for both groups.
Measure: Mean (Standard Deviation); unit: Global PSQI score
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 7 | 8
Global PSQI score
  Baseline | 4.714286 (1.799371) | 2.5 (1.414214)
  Day 28 | 4.571429 (4.117327) | 2.5 (1.85164)
  Day 72 | 4.125 (2.10017) | 1.88889 (1.536591)

ADVERSE EVENTS:
Time Frame: total 100 days for both interventions
Description: All adverse events, however minor, were documented in the CRF whether or not the Investigator concludes the event to be related to drug treatment. from baseline to end of trial visit.
Groups:
- Arm 1 Dolutegravir: Dolutegravir first - 50 mg once daily, day 0 to 44 (including a 2 week wash out period)
- Arm 1 No treatment: No treatment 28 days of the study, day 44 to 100
- Arm 2 No treatment: No treatment for the first 28 days of the study day 0 to 44
- Arm 2 Dolutegravir: Dolutegravir - 50 mg once daily, orally administered, day 44 to 100 (including a 2 week wash out period)
Arm/Group | Arm 1 Dolutegravir | Arm 1 No treatment | Arm 2 No treatment | Arm 2 Dolutegravir
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 1/8 | 0/8
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 8/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Dolutegravir (N=7) | Arm 1 No treatment (N=7) | Arm 2 No treatment (N=8) | Arm 2 Dolutegravir (N=8)
Transverse tibial metaphyseal (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Dolutegravir (N=7) | Arm 1 No treatment (N=7) | Arm 2 No treatment (N=8) | Arm 2 Dolutegravir (N=8)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hay fever (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cold (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Contact dermatitis on left ring finger (redness) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hit right cheek by cricket ball, swelling only (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5) | 5 (7) | 5 (6) | 5 (7)
low white blood cell count (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
low neutrophil count (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
low lymphocyte count (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
low monocyte (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
left wisdom tooth extraction because of decay and pain (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vivid Dreams (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep deprivation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Possible vasovagal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT04771754/Prot_SAP_000.pdf